CLINICAL TRIAL: NCT07189845
Title: Effect of Bispectral Index (BIS)-Guided Anesthesia on Postoperative Nausea and Vomiting in Children Aged 3 to 8 Years: A Prospective Randomized Controlled Trial
Brief Title: Effect of BIS-Guided Anesthesia on Postoperative Nausea and Vomiting in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Engin Çetin (Other Government)
Responsible Party: Sponsor-Investigator, Engin Çetin, principal investigator, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KSH-ANREA-EC-04
Record Dates: First submitted 2025-09-02; First posted 2025-09-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: PONV; BIS
Keywords: ponv; bıs
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIS GROUP (Active Comparator): BIS monitoring will be visible, and anesthesia depth will be adjusted according to BIS values (40-60).
  Interventions: Diagnostic Test: BIS GROUP
- CONTROL GROUP (Active Comparator): In the control group, the BIS monitor will be applied with the screen concealed from the investigator, and anesthesia depth will be guided solely by clinical parameters
  Interventions: Diagnostic Test: CONTROL GROUP

INTERVENTIONS:
Diagnostic Test: BIS GROUP — In the BIS group, monitoring will be visible and anesthesia depth will be maintained within a BIS value range of 40-60.
  Arms: BIS GROUP
Diagnostic Test: CONTROL GROUP — In the control group, the BIS monitor will be applied with the screen concealed from the investigator, and anesthesia depth will be guided solely by clinical parameters.
  Arms: CONTROL GROUP

SUMMARY:
This randomized controlled trial will evaluate the effect of bispectral index (BIS)-guided anesthesia on postoperative nausea and vomiting (PONV) in children aged 3-8 years undergoing elective adenoidectomy. Fifty-eight patients will be randomized to BIS-guided anesthesia (target 40-60) or standard clinical management. The primary outcome is PONV incidence within 24 hours. Secondary outcomes include antiemetic use, emergence time, hospital stay, and parental satisfaction.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind controlled trial aims to evaluate the effect of bispectral index (BIS)-guided anesthesia on postoperative nausea and vomiting (PONV) in children aged 3 to 8 years undergoing elective adenoidectomy. PONV is a common postoperative complication in pediatric surgery, with reported incidences of 30-70%, leading to delayed oral intake, prolonged hospital stay, and reduced parental satisfaction. BIS monitoring provides an objective EEG-based measure of anesthesia depth, allowing precise titration of anesthetic agents and potentially reducing postoperative complications. While adult studies and meta-analyses have shown that BIS guidance decreases the incidence of PONV, evidence in pediatric populations remains limited. A total of 58 ASA I-II patients will be randomized into two groups: BIS-guided anesthesia (target 40-60) and standard clinical parameter-guided anesthesia with the BIS screen hidden. The primary outcome is the incidence of PONV within 24 hours postoperatively. Secondary outcomes include antiemetic use, severity of PONV, time to emergence, length of hospital stay, and parental satisfaction assessed with a Likert scale. The findings of this trial are expected to clarify the role of BIS monitoring in improving postoperative outcomes in pediatric anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-8 years
* ASA physical status class I-II
* Scheduled for elective adenoidectomy
* Written informed consent obtained from parents

Exclusion Criteria:

* Children with a previous history of PONV
* Patients receiving antiemetic, steroid, or sedative medication
* Acute upper respiratory tract infection
* History of neurological or psychiatric disorders
* Body mass index (BMI) below the 5th percentile or above the 95th percentile
* Anatomical airway abnormalities

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) during the first 24 hours postoperatively. | T1: Immediately before extubation T2: 6 hours after extubation T3: 12 hours after extubation T4: 24 hours after extubation
  PONV will be assessed at postoperative intervals of 0-6, 6-12, and 12-24 hours. The Postoperative nausea and vomiting (PONV) will be assessed at postoperative intervals of 0-6, 6-12, and 12-24 hours. PONV severity will be evaluated using a predefined four-point ordinal scale based on the presence and frequency of nausea and vomiting, as follows:
  0: No nausea or vomiting
  1. Mild nausea
  2. Severe nausea or a single vomiting episode
  3. Severe nausea with multiple vomiting episodes or intractable PONV

SECONDARY OUTCOMES:
Emergence Time | From discontinuation of sevoflurane at the end of surgery until eye opening in response to verbal command, assessed up to 30 minutes
  Emergence time (defined as the time from discontinuation of sevoflurane until the patient opens their eyes in response to verbal command)
Antiemetic use and timing | 0-24 hours postoperatively
  The administration of rescue antiemetic drugs will be recorded for each patient within the first 24 hours after surgery. The specific agent used (e.g., ondansetron, dexamethasone), the time of administration, and the number of doses will be documented from anesthesia and nursing records. The outcome will be expressed as the proportion of patients requiring antiemetic medication and the mean time to first administration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frelich M, Sklienka P, Romanova T, Nemcova S, Bilena M, Strakova H, Lecbychova K, Jor O, Formanek M, Bursa F. The effect of BIS-guided anaesthesia on the incidence of postoperative nausea and vomiting in children: a prospective randomized double-blind study. BMC Anesthesiol. 2024 Jul 9;24(1):228. doi: 10.1186/s12871-024-02610-w. PMID 38982400